CLINICAL TRIAL: NCT05266924
Title: A Randomized, Parallel-group, Multi-Center, Assessor-blind Phase 3 Study to Compare the Efficacy, Safety and Ease of Use of Two Follicle Stimulating Hormone -Human Recombinant (r-hFSH) 900 IU (66.0 μg) / 1.5mL Solution for Injection in Prefilled Pen (Foligraf®- Manufactured by BSV and Gonal-f® Manufactured by Merck Serono) in Subjects Undergoing Controlled Ovarian Stimulation for Assisted Reproductive Technology
Brief Title: Recombinant Follicle-stimulating Hormone in Treatment for Infertility
Acronym: REFRESH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bharat Serums and Vaccines Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSV_rhFSH_20_09
Record Dates: First submitted 2022-01-23; First posted 2022-03-04 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Solutions; Injections; follitropin alfa

STUDY DESIGN:
Intervention Model Description: This is a Randomized, Parallel-group, Multi-Center, Assessor-blind Phase 3 Study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor including the investigator, outcoume assessor (sonography, embyrologist) shall be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Foligraf 900 IU (66.0 μg) / 1.5mL Solution for Injection in Prefilled Pen Follicle Stimulating Hormone (Human Recombinant) manufactured by Bharat Serums and Vaccines Ltd
  Interventions: Drug: Recombinant Human Follicle Stimulating Hormone 900 IU (66.0 μg) / 1.5mL Solution for Injection in Prefilled Pen
- Reference group (Active Comparator): Gonal-f Recombinant Human Follicle Stimulating Hormone
  Interventions: Drug: Recombinant Human Follicle Stimulating Hormone 900 IU (66.0 μg) / 1.5mL Solution for Injection in Prefilled Pen

INTERVENTIONS:
Drug: Recombinant Human Follicle Stimulating Hormone 900 IU (66.0 μg) / 1.5mL Solution for Injection in Prefilled Pen — fixed-dose of 225 IU/day, subcutaneous (SC), daily, for 5 days. further dosage will be adjusted till adequate follicular development.
  Other Names: Foligraf; Gonal-f

SUMMARY:
This is a randomized multi-centre, assessor-blind, parallel-group study to be conducted in 250 women in the age group of 20 to 39 years (both inclusive), who are indicated to undergo COS as part of assisted reproductive technology (ART). The participant will receive r-hFSH, fixed-dose for 5 days, and day 6 onwards the dose may be adjusted for a single cycle of COS followed by ART procedures, and post-ART follow-up for ongoing pregnancy.

The primary and secondary outcomes will be captured on days as per protocol. Adverse events will be noted for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has indication ART using COS.
* Subject has regular menstrual cycle of 21-35 days.
* Subject has one of the following:

  1. FSH level <10 IU/L and Estradiol levl <80 pg/mL at day 2 or 3
  2. Anti-mullerian hormone (AMH) level between 1 to 3.5 ng/mL during the menstrual cycle
* Subject has an antral follicle count (AFC) of 10- 25, follicle ≤10 mm in diameter before ovarian stimulation
* Subject has a BMI ≥18 and <30 kg/m2
* Subject has results of clinical laboratory tests within normal reference range
* Subject and her partner are willing to provide written informed consent and comply

Exclusion Criteria Details Subject has history of >2 failed ART cycles

* Subject with history of any endocrine abnormality, with documented hormone levels outside the reference range, which are clinically relevant, at screening
* Subject with a history of ovarian hyper-response (i.e., previous COS cycle with >25 follicles of ≥11 mm in diameter on USG) or OHSS
* Subject with documented polycystic ovarian syndrome (PCOS) at the time of screening
* Subject with only one ovary or ovarian abnormality (including endometrioma >10 mm; visible on USG), at screening
* Subject with documented severe endometriosis (American Society of Reproductive Medicine stage 3 or stage 4) or hydrosalpinx, at screening
* Subject with submucosal fibroids ≥5 cm or any other clinically relevant pathology, which could impair embryo implantation or pregnancy continuation, at screening
* Subject with a history of extrauterine pregnancy within 3 months of screening
* Subject with history of poor response to gonadotropin treatment (retrieval of <4 oocytes) in the previous ART cycle
* Subject with history of ≥3 miscarriages, at any time prior to screening
* Subject who has tested positive for Human Immunodeficiency Virus, Hepatitis B or Hepatitis C at screening
* Subject known to be allergic, hypersensitive, or intolerant to any of the preparations of r hFSH or its excipients, that will be used in the study
* Subject with contraindications to the use of gonadotropins (e.g., tumours, undiagnosed vaginal bleeding, or ovarian cysts) or gonadotropin-releasing hormone (GnRH) antagonists
* Subject with a history of epilepsy, thrombophilia, cardiovascular, gastrointestinal, hepatic, renal, pulmonary, auto-immune disease, or any active infection, requiring treatment which at the investigator's discretion might interfere with the study
* Subject with history of malignancy
* Subject who smokes or has stopped smoking within the last 3 months prior to screening
* Subject with history of alcohol or drug abuse within 12 months prior to screening
* Subject who has received any treatment listed below within 5 half-lives prior to screening:

  1. Any agent(s) known to affect ovulation (e.g., neuroleptics);
  2. Drugs known or suspected to be teratogenic in nature.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 250 (Estimated)
Dates: Start 2022-07-23 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | Oocyte pick up - up to ~ 34 to 36 hours after human chorionic gonadotropin (hCG) administration
  Number of oocytes retrieved

SECONDARY OUTCOMES:
Clinical pregnancy rate | 4 weeks after embryo transfer (ET)
  Clinical pregnancy rate
Ongoing Pregnancy rate | 11±1 weeks after ET
  Ongoing pregnancy rate
Cycle cancellation rate | at Stimulation phase up to 20 days, oocyte pick up up to ~ 34 to 36 hours after hCG administration, ET anytime up to 8 weeks
  Cycle cancellation rate
Total Doseof r-hFSH | at end of stimulation up to 20 days
  Total dose of r-hFSH (in IU) required for ovarian stimulation;
Number of Days of r-hFSH stimulation | at end of stimulation up to 20 days
  Number of days of r-hFSH stimulation
Number of subject Change in Dosage | post Day 6 till end of stimulation up to 20 days
  Proportion of subjects requiring change in dose
Hormonal Investigation | Day 6
  Estradiol, Luteinizing, Progesterone, and inhibin b levels
Follicle size on Day 6 | Day 6
  Number of follicles with size <11mm, Number of follicles with size 11- 14 mm, Number of follicles with size15 mm, Number of follicles with size16 mm, Number of follicles with size17 mm and Number of follicles with size ≥18 mm
Follicle size at HCG administration | Day of hCG administration anytime upto 3 weeks
  Number of follicles with size <11mm, Number of follicles with size 11- 14 mm, Number of follicles with size15 mm, Number of follicles with size16 mm, Number of follicles with size17 mm and Number of follicles with size ≥18 mm mm)
Endometrium thickness | day 6
  Endometrial thickness (mm)
Endometrium at HCG administration | day of hCG injection (anytime upto 3 weeks)
  Endometrial thickness (mm)
Number of Matured oocytes | Oocyte pick up ~ 34 to 36 hours after hCG administration
  Proportion of matured oocytes
Number of good quality embryos | ET day (up to 8 weeks)
  Number of good quality embryos
Number of Adverse events | Baseline, 1st day of stimulation, day 6 , end of stimulation up to 20 days, hCG administration, oocyte pick up ~ 34 to 36 hours after hCG administration, ET up to 8 weeks, clinical pregnancy (after 4 weeks of ET), ~12 weeks after ET
  Number of treatment-emergent adverse events (TEAE) reported
Specific adverse events | Day 1 of Stimulation till ~12 weeks after ET
  The number of patients with ovarian hyperstimulation syndrome (OHSS) reported
Exploratory | End of stimulation up to 20 days
  Ease of use of Pen - comparison of total score of Questionnaire to user of rhFSH pen
Evaluation of immunogenicity (antibody) of r-hFSH | Baseline, 4 weeks and 12 weeks
  Evaluation of immunogenicity of r-hFSH, comparison of antibody titre against r-hFSH in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Om Research Center Om Surgical Center and Maternity Home, Varanasi, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No